CLINICAL TRIAL: NCT02104635
Title: Postpartum Empowerment: an Integrated Approach Driving Demand and Delivery of High Quality, Low-cost Postnatal Services in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Jessica Cohen, Harvard School of Public Health (Unknown); Saving Lives at Birth Initiative (Unknown); Jacaranda Health (Other)
Responsible Party: Principal Investigator, Margaret McConnell, Assistant Professor of Global Health Economics, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Factorial | Purpose: Basic Science
Other Study IDs: Saving Lives at Birth
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Maternal and Newborn Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): The control group receives standard of care from Jacaranda clinic and does not receive any additional post-partum check-in from a community health worker.
- CHW-Visit (Experimental): The CHW-Visit group will receive a visit at their home from a community health worker (CHW) three days after delivery. The CHW will administer a checklist designed to identify maternal and newborn complications and will provide information about positive maternal health and care behaviors. The CHW will encourage women to return to the clinic at 7 days to receive a well-baby check.
  Interventions: Behavioral: Delivery of a Post-Partum Package
- CHW-Phone (Experimental): The CHW-Visit group will receive a phone call from a community health worker (CHW) three days after delivery. The CHW will administer a checklist designed to identify maternal and newborn complications and will provide information about positive maternal health and care behaviors. The CHW will encourage women to return to the clinic at 7 days to receive a well-baby check.
  Interventions: Behavioral: Delivery of a Post-Partum Package

INTERVENTIONS:
Behavioral: Delivery of a Post-Partum Package
  Arms: CHW-Phone; CHW-Visit

SUMMARY:
This research represents a randomized trial of a program to improve timely postnatal care, comparing post-natal check-ups performed by community health workers delivered either by phone or in person to a control group. The study hypothesis is that when community health workers check on women three days after their delivery we will see improvements in the detection of maternal and child complications, better knowledge of complications and an increase in behaviors that are expected to lead to improved maternal and child health.

ELIGIBILITY:
Inclusion Criteria:

Women between 18 and 40 years old are eligible for inclusion if they have had a safe normal delivery of a live infant delivery at a Jacaranda Health facility. Eligible women must reside in a 20 km radius from the Jacaranda Health's hospital facility in peri-urban Nairobi. Women must provide a phone number to where they expect that can be reached 2 weeks postpartum.

Exclusion Criteria:

Women who elect to leave the Jacaranda Health facility before the recommended 24 hours, against medical advice, postpartum are not eligible to participate in the postpartum care study. Women and their newborns who are referred to another hospital for higher level emergency obstetric or neonatal care will not be eligible to participate. Women who relocate outside the defined geographic area surrounding the hospital after their delivery are also not eligible.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Enrollment: 109 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Complications detected | 3 days after delivery
  Any maternal complications detected Number of maternal complications detected Any newborn complications detected Number of newborn complications detected
Successful referrals | 10 days after delivery (survey and administrative records)
  If CHW made referral on day 3 for baby, respondent went to health facility If CHW made referral on day 3 for mother, respondent went to health facility
Care Seeking Behavior around complications and well baby check-up | 10 days after delivery (survey)
  Brought baby to health facility for a well-baby check up If maternal complications (self-reported) in past week, visited or called health facility If baby complications (self-reported) in past week, visited or called health facility
Knowledge of danger signs | 10 days after delivery (survey)
  Can name any maternal danger signs for which care should be sought (at day 10) Number of maternal danger signs named for which care should be sought (at day 10). Note: if mother lists "other" danger signs not coded, these should be coded as appropriate danger signs for which care should be sought or not Can name any baby danger signs for which care should be sought (at day 10) Number of baby danger signs named for which care should be sought (at day 10). Note: if mother lists "other" danger signs not coded, these should be coded as appropriate danger signs for which care should be sought or not
Breastfeeding | 10 days and 9 weeks after delivery (survey)
  Fed only breastmilk in past week

SECONDARY OUTCOMES:
Referrals | 3 days after delivery (from admin records)
  Any referral made for mother Any referral made for newborn
Feeding behavior | 10 days 9 week after delivery (survey)
  Fed baby at least 3 times in past 8 hours (at 10 days) Fed baby at least 2 times in past 8 hours (at 9 weeks) No complications breastfeeding in past week (at 10 days and at 9 weeks) Applied nothing/only water to umbilical stump (at 10 days) Ate any protein (at 10 days and at 9 weeks) Mentions keeping baby warm for bath (at 10 days) Feeds baby at night (at 10 days) Using any family planning method (at 9 weeks)
Care seeking regarding breastfeeding, vaccines and child wellness | 10 days and 9 weeks after delivery (survey)
  If had complication breastfeeding, visited or called health facility (at day 10) Baby has had first vaccine course in a timely manner, should be at 6 weeks according to Kenyan recommendations (measured at 9 weeks) Baby was brought in for child wellness check up (measured at 9 weeks)
Knowledge of feeding and safety | 10 days after delivery (survey)
  Mentions feeding at least 3 times in 8 hours Knows two types of protein mother can eat Knows to keep baby warm while bathing Knows to feed baby at night Knows to keep cord clean and dry to prevent infection Knows to wash hands after going to toilet Knows to wash hands before touching/holding baby Knows to wash hands after changing diaper
Care seeking at Jacaranda Health | 10 days after delivery (survey)
  Brought baby to JH within 10 days of delivery for any reason Mother came to JH within 10 days of delivery for any reason Brought baby to JH within 10 days of delivery for well-baby visit

CONTACTS AND LOCATIONS:
Locations (1):
- Jacaranda Health, Nairobi, Kenya

REFERENCES:
- [Derived] McConnell M, Ettenger A, Rothschild CW, Muigai F, Cohen J. Can a community health worker administered postnatal checklist increase health-seeking behaviors and knowledge?: evidence from a randomized trial with a private maternity facility in Kiambu County, Kenya. BMC Pregnancy Childbirth. 2016 Jun 4;16(1):136. doi: 10.1186/s12884-016-0914-z. PMID 27260500